

# Minimal Opioid Use After Total Hip Replacement (THR): A Blinded, Randomized, Placebo-Controlled Study

FUNDER: Anesthesiology Department,

Hospital for Special Surgery

PROTOCOL NO.: 2017-0721

DATE: 0625/2020

This document contains the confidential information of the Hospital for Special Surgery. It is provided to you and your company's personnel for review. Your acceptance of this document constitutes an agreement that you will not disclose the information contained herein to others without the prior written consent of the Hospital for Special Surgery. No other use or reproduction is authorized by Hospital for Special Surgery, nor does the Hospital for Special Surgery assume any responsibility for unauthorized use of this protocol.




# **TABLE OF CONTENTS**

| | LE OF CONTENTS | |
|---|---|---|
| PRO | TOCOL SYNOPSIS | 3 |
| 1.0 | INTRODUCTION | |
| 2.0 | PRODUCT DESCRIPTION | |
| 3.0 | OBJECTIVE OF CLINICAL STUDY | 4 |
| 4.0 | STUDY HYPOTHESIS | 4 |
| 5.0 | STUDY DESIGN | 4 |
| 5.1 | Study Duration | 4 |
| 5.2 | Endpoints | 4 |
| 5.2 | 2.1 Primary Endpoint | 4 |
| 5.2 | 2.2 Secondary Endpoints | 4 |
| 5.2 | 2.3 Safety Evaluations | 4 |
| 5.3 | Study Site | |
| 6.0 | STUDY POPULATION | 4 |
| 6.1 | Number of Subjects | 4 |
| 6.2 | Inclusion Criteria | |
| 6.3 | Exclusion Criteria: | |
| 6.4 | Randomization | |
| 7.0 | PROCEDURES | - |
| 7.1 | Surgical Procedure | |
| | 1.1. Investigational Product Administration | |
| 7.2 | Imaging Procedure | |
| 7.3 | Medical Record Requirements | |
| 7.4 | Data Collection | |
| 7.5 | Schedule of Assessments | |
| 7.6 | Radiological Evaluations | |
| 7.7 | Clinical Evaluations | |
| | 7.1. Revision Surgery | |
| 8.0 | STATISTICAL ANALYSIS | |
| 9.0 | ADVERSE EVENT ASSESSMENT | |
| 9.1 | Adverse Event (AE) | |
| 9.2 | Serious Adverse Events (SAE) | |
| 9.3 | Subsequent Surgical Interventions Definitions | |
| 9.4 | Adverse Event Relationship | |
| 9.5 | Adverse Event Recording | |
| 9.6<br><b>10.0</b> | Adverse Event Reporting INVESTIGATOR RESPONSIBILITIES, RECORD AND REPORTS | |
| 10.0 | Subject Consent and Information | |
| 10.1 | · | |
| 10.2 | - · · <b>,</b> - · | |
| 10.3 | | |
| 10.4 | | |
| 10.5 | 3 | |
| 11.0 | REFERENCES | |
| _ | ENDIX A: Case Report Forms | |
| | | 🧸 |



# **PROTOCOL SYNOPSIS**

| Protocol Title: | Minimal Opioid use after Total Hip Replacement (THR): a blinded randomized placebo-controlled study |
|---|---|
| Protocol Number: | 2017-0721 |
| Protocol Date: | 6/25/2020 |
| Sponsor: | Hospital for Special Surgery, Department of Anesthesiology |
| Principal Investigator: | Kethy Jules-Elysee, MD |
| Objective: | Total hip arthroplasty can be associated with significant postoperative pain. Side effects of pain management may impair participation in physical therapy and slow readiness for discharge from the hospital. In a previous study done by our group, epidural patient-controlled analgesia (EPCA) with a hydromorphone containing solution appeared to have a more favorable pain profile with ambulation, but greater side effects compared to injection of a peri-articular cocktail. The use of opioid was greater in the peri-articular injection group (PAI). There was no difference in length of stay. In view of the controversy over opioid use, we would like to develop an optimal opioid sparing pain management approach by comparing 3 different protocols 1) Plain local anesthetic EPCA; 2) PAI; 3) EPCA + PAI; all in conjunction with a multimodal opioid sparing pain regimen. The goal would be to maximize pain control while minimizing opioid use and side-effects. |
| Study Design: | Randomized Controlled Clinical Trial |
| Enrollment: | 180 total (60 in each group) |
| Subject Criteria: | <ul> <li>Patients with osteoarthritis scheduled for primary total hip arthroplasty with participating surgeon</li> <li>Age 45 to 80 years old</li> <li>Planned use of regional anesthesia</li> <li>Ability to follow study protocol</li> <li>Planned posterolateral surgical approach</li> </ul> |
| Study Duration: | Enrollment Period: Pre-op, intra-op, post-op (POD0-3, 7, 90);<br>Duration of Follow ups: Approximately 15 mins each |
| Data Collection: | Collected from medical records and patient. |
| Outcome<br>Parameters: | <ul> <li>Opioid use (oral morphine equivalents, cumulative, within<br/>24 hours).</li> </ul> |




#### 1.0 INTRODUCTION

Total hip arthroplasty can be associated with significant postoperative pain. Side effects of pain management may impair participation in physical therapy and slow readiness for discharge from the hospital. In a previous study done by our group, epidural patient controlled analgesia (EPCA) with a hydromorphone containing solution appeared to have a more favorable pain profile with ambulation, but greater side effects compared to injection of a peri-articular cocktail. The use of opioid was greater in the peri-articular injection group (PAI). There was no difference in length of stay. In view of the controversy over opioid use, we would like to develop an optimal opioid sparing pain management approach by comparing 3 different protocols 1) Plain local anesthetic EPCA; 2) PAI; 3) EPCA + PAI; all in conjunction with a multimodal opioid sparing pain regimen.

# 2.0 OBJECTIVE OF CLINICAL STUDY

The objective of this study is to maximize pain control while minimizing opioid use and side effects.

#### 3.0 STUDY HYPOTHESES

Hypothesis 1: Compared to EPCA or PAI alone, the EPCA + PAI protocol will result in:

- lower opioid utilization
- lower pain scores
- lower opioid-related symptom distress scales
- improved quality of recovery scores
- higher patient satisfaction.

<u>Hypothesis 2:</u> The use of EPCA + PAI protocol will lead to earlier "readiness for discharge" to home or to a rehab facility compared to plain EPCA alone or PAI alone.

#### 4.0 STUDY DESIGN

# 4.1 Endpoints

# 4.1.1 Primary Endpoint

Opioid use (oral morphine equivalents, cumulative, within 24 hours).

# 4.1.2 Secondary Endpoints

- Pain at rest via NRS scale (POD 1,2,3, until D/C POD7 and 90)
- Pain with physical therapy via NRS scale (POD 1,2,3,until D/C POD7 and 90)
- Opioid side effects via ORSDS guestionnaire (POD1,2)
- Post-operative pain via Pain OUT questionnaire (POD 1)




- Patient satisfaction (0-10 Likert scale) regarding pain control (POD 1, 2, 3; POD7 & POD90)
- Neuropathic pain via S-LANSS SF-8 (Pre-Op, POD 7 & 90)
- Quality of Recovery via QoR-40 (POD 1,2,3)
- Readiness for discharge time (At D/C)

# 4.2 Study Sites

This study will take place at the main campus of the Hospital for Special Surgery.

# 5.0 STUDY POPULATION

# 5.1 Number of Subjects

180 subjects (60 in each group).

#### 5.2 Inclusion Criteria

Subjects of either gender will be included if:

- Patients with osteoarthritis scheduled for primary total hip arthroplasty with participating surgeon
- Age 45 to 80 years old
- Planned use of regional anesthesia
- Ability to follow study protocol
- Planned posterolateral surgical approach

#### 5.3 Exclusion Criteria

Subjects will be excluded from the study if:

- Patients younger than 45 years old and older than 80
- Patients intending to receive general anesthesia
- Patients with an ASA of IV
- Patients with insulin-dependent diabetes
- Patients with hepatic (liver) failure (history of cirrhosis or elevated LFT's)
- Patients with chronic renal (kidney) failure (formal diagnosis of renal disease of elevated creatinine)
- Chronic opioid use (taking opioids for longer than 3 months on a daily basis)
- Patients with any prior major ipsilateral hip surgery

#### 5.4 Randomization

A block randomization scheme will be created by a statistician not involved with the study. Prior to study start, 1) the randomization scheme will be shared with pharmacy, and 2) sealed envelopes containing only the PAI portion of the randomization assignments will be prepared by an unaffiliated RA and attached to the study enrollment folders. When a patient is enrolled, pharmacy will be notified and they will prepare the EPCA solution according to the randomization scheme. The sealed envelope will be given to the physician who will open




it to reveal the PAI portion of the randomization. This way the anesthesiologist and surgeon can remain blinded as to the EPCA (active vs. placebo) portion of the randomization.

# 6.0 PROCEDURES

# 6.1 Surgical Procedure

# **EPCA GROUP**

# Pre-Operative Anesthesia/Analgesia

- Baby ASA 81 mg
- Cymbalta 60mg
- Clonidine Patch 0.1mg for 24hr

# **Operating Room**

- Anesthetic: Combined Spinal-Epidural with 1.5% Mepivacaine (4 cc), (if need to induce hypotension, give Mepivacaine through epidural). IV sedation with Midazolam, Propofol (no opioids) \*Ketamine 20 mg prior to incision 30 mg in Propofol infusion
- IV TXA 10 mg/kg up to 1000mg
- Antiemetic: 20mg famotidine (Pepcid) and 4mg ondansetron (Zofran) + \*8 mg IV Decadron
- \*IV Tylenol prior to transfer to PACU
- End of case: \*Toradol (Ketorolac) (30 mg IV if age 64 or younger, 15 mg IV if age >=65 or weight <50 kg)</li>

#### **Post-Operative Procedures**

- Foley catheter until POD 1 at 10:00 AM. Oral diet and physical therapy upon block resolution.
- Cymbalta 60 mg qd POD1-2
- PCEA (Bupivacaine 0.06%) (4/4/10/20, initially).
- Reduce PCA (0/4/10/20 POD1, 6:59). D/C PCA (POD1, 10:00)
- Ondansetron (IV 4 mg q 8 hr PRN)
- Nalbuphine (IV 5 mg g 6 hr PRN)
- Continue IV Acetaminophen (1000 mg q 6 hr for 3 doses followed by oral dosing q 6hr)
- Toradol (30 mg IV g 6 hr until POD 1, total 4 doses including OR dose)
- Oxycodone (5 mg q 3 hr PRN for mild pain / 10 mg for moderate to severe pain)
- Celebrex 200 mg bid on POD 1
- IV Pepcid 20 mg g 12 hr
- Dilaudid (1 mg SQ q 4 hr PRN, after PCA D/C)
- Remove Clonidine Patch 24 hours after application
- Miralax 17g daily
- ASA 325mg bid

# PAI GROUP




# Pre-Operative Anesthesia/Analgesia

- Baby ASA 81 mg
- Cymbalta 60mg
- Clonidine Patch 0.1mg for 24hr

# **Operating Room**

- A. <u>Anesthetic:</u> At end of surgery, the surgeon performs a peri-articular injection. Protocolized method for injection. \*Deep Injection: (0.5% Bupivacaine with Epi, 30ml; morphine, 8 mg/ml, 1ml; methylprednisolone, 40 mg/ml, 1ml; cefazolin, 500 mg in 10 ml; normal saline, 22ml). Superficial injection: (40 ml 0.25% Bupivacaine).
- B. <u>Anesthetic:</u> Combined Spinal-Epidural with 1.5% Mepivacaine (4 cc) (if needed, can add lidocaine to epidural), (if need to induce hypotension, give Mepivacaine through epidural). IV sedation with Midazolam, Propofol (no opioids) \*Ketamine 20 mg prior to incision 30 mg in Propofol infusion
- IV TXA 10 mg/kg up to 1000mg
- <u>Antiemetic</u>: 20mg famotidine (Pepcid) and 4mg ondansetron (Zofran).\*No Decadron because of steroids in injection.
- \*IV Tylenol 1000 mg prior to transfer to PACU
- End of case: \*Toradol (Ketorolac) (30 mg IV if age 64 or younger, 15 mg IV if age >=65 or weight <50 kg)</li>

#### **Post-Operative Procedures**

- Foley catheter until POD 1 at 10:00 AM. Oral diet and physical therapy upon block resolution.
- Cymbalta 60 mg qd POD1-2
- Placebo epidural pain pump containing normal saline, programmed as such:
   4/4/10/20, initially. Reduce PCA (0/4/10/20 POD 1, 6:59). D/C PCA (POD 1 10:00)
- Ondansetron (IV 4 mg q 8 hr PRN)
- Nalbuphine (IV 5 mg g 6 hr PRN).
- Continue IV Acetaminophen (1000 mg q 6 hr for 3 more doses following oral dosing q 6 hr)
- Toradol (30 mg q 6 hr until POD 1, total 4 doses including OR dose)
- Oxycodone q 3 hr PRN (5 mg for mild pain / 10 mg for moderate to severe pain)
- Celebrex 200 mg bid on POD 1
- IV Pepcid 20 mg q 12hr
- Dilaudid (1 mg SQ q 4 hr PRN, after PCA discontinuation)
- Remove Clonidine Patch 24 hours after application
- Miralax 17g daily
- ASA 325 mg bid

#### EPCA + PAI GROUP

# Pre-Operative Anesthesia/Analgesia

- Baby ASA 81 mg
- Cymbalta 60mg
- · Clonidine Patch 0.1mg for 24hr

# **Operating Room**






- <u>Anesthetic</u>: Combined Spinal-Epidural with 1.5% Mepivacaine (4 cc), (if need to induce hypotension, give Mepivacaine through epidural). IV sedation with Midazolam, Propofol (no opioids) \*Ketamine 20 mg prior to incision 30 mg in Propofol infusion
- IV TXA 10 mg/kg up to 1000mg
- Antiemetic: 20mg famotidine (Pepcid) and 4mg ondansetron (Zofran)
- \*IV Tylenol prior to transfer to PACU
- End of case: \*Toradol (Ketorolac) (30 mg IV if age 64 or younger, 15 mg IV if age >=65 or weight <50 kg)</li>
- \*No Decadron given
- C. At end of surgery, the surgeon performs a peri-articular injection. Protocolized method for injection. \*Deep Injection: (0.5% Bupivacaine with Epi, 30ml; morphine, 8 mg/ml, 1ml; methylprednisolone, 40 mg/ml, 1ml; cefazolin, 500 mg in 10 ml; normal saline, 22ml). Superficial injection: (40 ml 0.25% Bupivacaine).

#### **Post-Operative Procedures**

- Foley catheter until POD 1 at 10:00 AM. 3. Oral diet and physical therapy upon block resolution.
- Cymbalta 60 mg qd POD1-2
- PCEA (Bupivacaine 0.06%) (4/4/10/20, initially).
- Reduce PCA (0/4/10/20 POD1, 6:59). D/C PCA (POD1, 10:00)
- Ondansetron (IV 4 mg q 8 hr PRN)
- Nalbuphine (IV 5 mg q 6 hr PRN)
- Continue IV Acetaminophen (1000 mg q 6 hr for 3 doses followed by oral dosing q 6hr)
- Toradol (If age <=64, 30 mg IV q 6 hr until POD 1, total 4 doses including OR dose)</li>
   If age >=65 or weight <50kg, 15mg</li>
- Oxycodone (5 mg q 3 hr PRN for mild pain / 10 mg for moderate to severe pain)
- Celebrex 200 mg bid on POD 1
- IV Pepcid 20 mg g 12 hr
- Dilaudid (1 mg SQ g 4 hr PRN, after PCA D/C)
- Remove Clonidine Patch 24 hours after application
- Miralax 17g daily
- ASA 325mg bid

#### 6.2 Data Collection

Data will be collected by an investigator or research assistant. Sources of data include medical records and patient physical assessments/interviews conducted by study personnel. Data will be recorded and managed using REDCap electronic data capture tools hosted at the Clinical and Translational Science Center (CTSC) at Weill Cornell Medical College. REDCap (Research Electronic Data Capture) is a secure, web-based application designed to support data capture for research studies, providing: 1) an intuitive interface for validated data entry; 2) audit trails for tracking data manipulation and export procedures; 3) automated export procedures for seamless data downloads to common statistical packages; and 4) procedures for importing data from external sources. Connection to REDCap occurs via the




hospital's encrypted cable and wireless networks, and data will be entered through a password protected computer terminal or iPad.

# The following data will be collected:

# Pre-operative/Baseline

- basic demographic data
- patient weight & height, BMI
- Comorbidities
- NRS Pain score at rest and with activity
- SF-8 Acute
- S-LANSS

#### POD 1

- date of surgery
- type of surgery
- NRS pain score at rest and with activity
- ORSDS
- QoR-40
- Pain outcomes questionnaire
- Opioid dose
- Patient Satisfaction

# POD 2

- NRS pain score at rest and with activity
- ORSDS
- QoR-40
- Opioid dose
- Patient satisfaction

#### POD 3

- NRS pain score at rest and with activity
- QoR-40
- Opioid dose
- Patient satisfaction

# At Discharge

Blinding assessment

# POD 7 (Phone F/U)

- NRS pain score at rest and with activity
- SF-8 Acute
- S-LANSS
- Blinding Assessment
- Opioid dose
- Patient satisfaction






# 90 Days (Phone F/U)

- NRS pain score at rest and with activity
- SF-8 Acute
- S-LANSS
- Opioid dose
- Patient satisfaction


# 6.3 Schedule of Assessments

| Procedures | Role | Day<br>Before<br>Surgery | Pre-Op | POD1 | POD2 | POD3 | At<br>Discharge | POD 7 | 90 Day<br>Phone<br>F/U |
|---|---|---|---|---|---|---|---|---|---|
| Eligibility Review | RA | Х | | | | | | | |
| Obtain Consent | Anes MD<br>or RA | | Х | | | | | | |
| Demographics | RA | | Х | | | | | | |
| Comorbidities | RA | | Х | | | | | | |
| NRS Pain at rest/with activity | RA | | Х | Х | Х | Х | | Χ | Χ |
| SF-8 Acute | RA | | Х | | | | | Х | Х |
| S-LANSS | RA | | Х | | | | | Х | Х |
| ORSDS | RA | | | Х | Х | | | | |
| QoR-40 | RA | | | Х | Х | Χ | | | |
| Pain Outcomes | RA | | | Х | | | | | |
| Questionnaire | | | | | | | | | |
| Blinding Assessment | RA | | | | | | Х | Х | |
| Opioid Dose | RA | | | Х | Х | Х | | Х | Х |
| Patient Satisfaction | RA | | | Х | Х | Х | | Х | Х |


# 7.0 STATISTICAL ANALYSIS

- Proposed analysis (e.g., student's t-test, ANOVA, chisquare, regression, etc.):
   Independent two sample t-tests
- Alpha level: 0.05/2 = 0.025. The primary goal of the study is to compare the
  combined intervention (EPCA+PAI) with EPCA alone and PAI alone. We ran a
  conservative power analysis for these two comparisons by applying Bonferroni
  corrections. We assume that EPCA alone and PAI alone will have similar effects.
  The comparison between these two groups is not the primary interest of the study.
- Beta or power level: 80%
- Primary outcome variable estimate (mean +/s.d. for continuous outcome): Mean ± SD opioid use (in 24hr)= 26 ± 22 mg OME
- Number of groups being compared (use 1 for paired analysis within the same subjects): 2 (assuming that there is no difference between EPCA alone and PAI alone).
- Effect size or change expected between groups: Opioid use (in 24hr): 50% reduction in OME
- Sample size: We would need 60 patients per group to achieve 80% power for detecting the above effect size for opioid use. The sample size accounts for 10% missing observations due to withdraws, losses to follow up, etc.

Continuous variables and discrete variables will be presented as mean+/-sd and proportion, respectively. Univariate analysis including t-test/Mann-Whitney Wilcoxon Rank test and Chisquare/Fisher's exact test will be conducted to compare continuous and discrete outcomes (both primary and secondary) between any two groups, respectively. Standard linear regression analysis can be used to compare opioid use between the intervention groups

#### 8.0 ADVERSE EVENT ASSESSMENT

All Adverse Events (AEs) will be reported in the final study report. Definitions for Adverse Event (AE) used in this study are listed below and are based on FDA and international guidelines:

# 8.1 Adverse Event Reporting

We will have data safety board to check if patients in the study experience increased pain, decreased quality of recovery and decreased satisfaction with the proposed regimens. The following physicians will be part of the safety board: Dr. Kirksey, Dr. DelPizzo, Dr. Memtsoudis.

# **Individual Stopping Criteria:**

The DSMB will review data related to the following individual stopping criteria:

- Gastrointestinal bleeding
- Hematoma






Blood in stool and/or vomit

Incidences of these potential issues will be reported to the IRB using the SAE

reporting form (attachment 3). The DSMB may recommend modification to individual stopping rules if necessary and may recommend stopping the study for the following reasons:

- The data show a significantly increased risk of serious adverse effects from the established incidence in the literature.
- If any mortality is seen in study participants
- All serious adverse events (SAE) will be reported within 5 days of the occurrence to the DSMB

#### 9.0 REFERENCES

- 1. Block BM, Liu SS, Rowlingson AJ, Cowan AR, Cowan JA Jr, Wu CL. Efficacy of Postoperative Epidural Analgesia: A Meta-analysis. JAMA 2003;290:2455-2463.
- 2. Ranawat AS and Ranawat CS. Pain management and accelerated rehabilitation for total hip and total knee arthroplasty. J Arthroplasty 2007;22:12-15.
- 3. Parvataneni HK, Shah VP, Howard H, Cole N, Ranawat AS, Ranawat CS. Controlling pain after total hip and knee arthroplasty using a multimodal protocol with local periarticular injections: A prospective randomized study. J Arthroplasty 2007;22:33-8.
- 4. Andersen KV, Pfeiffer-Jenses M, Haraldsted V, Soballe K. Reduced hospital stay and narcotic consumption, and improved mobilization with local and intraarticular infiltration after hip arthroplasty: a randomized clinical trial of an intraarticular technique versus epidural infusion in 80 patients. Acta Orthop 2007;78:180-6.
- 5. JulesElysee KM, Goon AK, Westrich GH, Padgett DE, Mayman DJ, Ranawat AS, Ranawat CS, Lin Y, Kahn RL, Bhagat DD, Goytizolo EA, Ma Y, Reid SC, Curren J, YaDeau JT. PatientControlled Epidural Analgesia or Multimodal Pain Regimen with Periarticular Injection After Total Hip Arthroplasty. J Bone Joint Surg Am, May 2015; 97 (10): 789798
- 6. Todd KH, Funk KG, Funk JP, et al. Clinical significance of reported changes in pain severity. Ann Emerg Med 1996; 27(4): 485–489
- 7. Alam A, Gomes T, Zheng H, Mamdani MM, Juurlink DN, Bell CM. Long-term analgesic use after low-risk surgery: a retrospective cohort study. Arch Intern Med. 2012 Mar 12;172(5):425-30
- 8. Rowe JW, Andres R, Tobin JD, Norris AH, Shock NW. The effect of age on creatinine clearance in men: a cross-sectional and longitudinal study. J Gerontol 1976 Mar;31(2):155-63.
- 9. Vestergaard P, Rejnmark L, Mosekilde L. Fracture risk associated with the use of morphine and opiates. J Intern Med. 2006 Jul;260(1):76-87.
- 10. Dowell D, Haegerich TM, Chou R. CDC Guideline for Prescribing Opioids for Chronic Pain--United States, 2016. JAMA. 2016 Apr 19;315(15):1624-45.
- 11. Clarke H, Soneji N, Ko DT, Yun L, Wijeysundera DN. Rates and risk factors for prolonged opioid use after major surgery: population based cohort study. BMJ. 2014 Feb 11;348:q1251.




12. YaDeau JT, Brummett\*CM, Mayman DJ, Lin Y, Goytizolo EA, Padgett DE, Alexiades MM, Kahn RL, Jules-Elysee KM, Westrich G, Gadulov Y, Fields KG, Goon AK,. Does Duloxetine Reduce Sub-Acute Pain After Knee Arthroplasty? A Randomized Controlled Trial. Best of Meeting: American Society of Regional Anesthesia and Pain Medicine. Feb 23, 2015.

13. Cuellar JM, Petrizzo A, Vaswani R, Goldstein, Bendo. Does Aspirin Administration Increase Perioperative Morbidity in Patients With Cardiac Stents Undergoing Spinal Surgery? Spine (Phila Pa 1976). 2015 May 1;40 (9):629-35.

- 14. Mantz J, Samama CM, Tubach F, et al. Impact of preoperative maintenance or interruption of aspirin on thrombotic and bleeding events after elective non-cardiac surgery: the multicentre, randomized, blinded, placebocontrolled, STRATAGEM trial. Br J Anaesth 2011;107:899–910
- 15. Chechik O, Thein R, Fichman G, et al. The effect of clopidogrel and aspirin on blood loss in hip fracture surgery. Injury 2011;42:1277–82
- 16. Morris T, Stables M, Hobbs A, de Souza P, Colville-Nash P, Warner T, Newson J, Bellingan G, Gilroy DW. Effects of Low-Dose Aspirin on Acute Inflammatory Responses in Humans. J Immunol, 2009 Aug 1;183(3):2089-96
- 17. Aspirin in patients undergoing non-cardiac surgery. Devereaux PJ, Mrkobrada M, Sessler DI, Leslie K, Alonso-Coello P, Kurz A, Villar JC, Sigamani A, Biccard BM, Meyhoff CS, Parlow JL, Guyatt G, Robinson A, Garg AX, Rodseth RN, Botto F, Lurati Buse G, Xavier D, Chan MT, Tiboni M, Cook D, Kumar PA, Forget P, Malaga G, Fleischmann E, Amir M, Eikelboom J, Mizera R, Torres D, Wang CY, VanHelder T, Paniagua P, Berwanger O, Srinathan S, Graham M, Pasin L, Le Manach Y, Gao P, Pogue J, Whitlock R, Lamy A, Kearon C, Baigent C, Chow C, Pettit S, Chrolavicius S, Yusuf S; POISE-2 Investigators. N Engl J Med. 2014 Apr 17;370(16):1494-50

